CLINICAL TRIAL: NCT01316900
Title: A Multicenter Trial Comparing the Efficacy and Safety of GSK573719/GW642444 With GW642444 and With Tiotropium Over 24 Weeks in Subjects With COPD
Brief Title: 24-week Trial Comparing GSK573719/GW642444 With GW642444 and With Tiotropium in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113360
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting muscarinic antagonist; tiotropium; COPD; long-acting beta agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; fluticasone furoate-vilanterol trifenatate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK573719/GW642444 125/25 (Experimental): 125/25 mcg once-daily
  Interventions: Drug: GSK573719/GW642444 125/25
- GSK573719/GW642444 62.5/25 (Experimental): 62.5/25 mcg once-daily
  Interventions: Drug: GSK573719/GW642444 62.5/25
- GW642444 (Experimental): 25 mcg once-daily
  Interventions: Drug: GW642444
- tiotropium bromide (Active Comparator): 18 mcg once-daily
  Interventions: Drug: tiotropium bromide

INTERVENTIONS:
Drug: GSK573719/GW642444 125/25 — 125/25 mcg once-daily
  Other Names: GSK573719/vilanterol trifenatate
  Arms: GSK573719/GW642444 125/25
Drug: GSK573719/GW642444 62.5/25 — 62.5/26 mcg once-daily
  Other Names: GSK573719/vilanterol trifenatate
  Arms: GSK573719/GW642444 62.5/25
Drug: GW642444 — 25 mcg once-daily
  Other Names: vilanterol trifenatate
  Arms: GW642444
Drug: tiotropium bromide — 18 mcg once-daily
  Arms: tiotropium bromide

SUMMARY:
This is a Phase III multicenter, randomized, double-blind, double-dummy, parallel-group study to evaluate the efficacy and safety of two doses of GSK573719/GW642444 Inhalation Powder and GW642444 Inhalation Powder via a Novel Dry Powder Inhaler and tiotropium via HandiHaler when administered once-daily over a 24-week treatment period in subjects with chronic obstructive pulmonary disease (COPD). Subjects who meet eligibility criteria at Screening (Visit 1) will complete a 7 to10 day run-in period followed by a randomization visit (Visit 2) then a 24-week treatment period. There will be a total of 9 clinic study visits. A follow-up phone contact for adverse event assessment will be conducted approximately one week after the last study visit (Visit 9 or Early Withdrawal). The total duration of subject participation in the study will be approximately 26 weeks. The primary measure of efficacy is clinic visit trough (pre-bronchodilator and pre-dose) forced expiratory volume in one second (FEV1) on Treatment Day 169. Safety will be assessed by adverse events, 12-lead ECGs, vital signs, and clinical laboratory tests.

DETAILED DESCRIPTION:
This is a 24-week, Phase III multicenter, randomized, double-blind, double-dummy, parallel-group study. Eligible subjects will be randomized to GSK573719/GW642444 125/25mcg, GSK573719/GW642444 62.5/25mcg, GW642444 25mcg, or tiotropium treatment groups in a 1:1:1:1 ratio. Treatments will be administered once-daily in the morning by inhalation using a Novel Dry Powder Inhaler (Novel DPI) and HandiHaler. There will be a total of 9 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 7 to 10 day run-in period followed by a 24-week treatment period. Clinic visits will be at Screening, Randomization (Day 1), Day 2, after 4, 8, 12, 16, and 24-weeks of treatment, and 1 day after the Week 24 Visit (also referred as Treatment Day 169). A follow-up contact for adverse assessment will be conducted by telephone approximately 7 days after Visit 9 or the Early Withdrawal Visit. The total duration of subject participation, including follow-up will be approximately 26 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the run-in and study treatment periods. At screening, pre-bronchodilator spirometry testing will be followed by post-albuterol/salbutamol spirometry testing. Post-albuterol/salbutamol FEV1 and FEV1/forced vital capacity (FVC) values will be used to determine subject eligibility. To further characterize bronchodilator responsiveness, post-ipratropium testing will be conducted following completion of post-albuterol/salbutamol spirometry. Spirometry will be conducted at each post-randomization clinic visit. Six hour post-dose serial spirometry will be conducted at Visits 2, 6, and 8. Trough spirometry will be obtained 23 and 24 hours after the previous day's dose of blinded study medication at Visits 3 to 9. All subjects will be provided with an electronic diary (eDiary) for completion daily in the morning and the evening throughout the run-in and treatment periods. Subjects will use the eDiary to record peak expiratory flow (PEF) each morning, dyspnea scores using the Shortness of Breath with Daily Activities instrument (SOBDA), daily use of supplemental albuterol/salbutamol as either puffs/day from a metered-dose inhaler (MDI) and/or nebules used per day, and any healthcare contacts related to COPD. Additional assessments of dyspnea will be obtained using the Baseline and Transition Dyspnea Index (BDI/TDI) which is an interviewer based instrument. At Visit 2, the severity of dyspnea at baseline will be assessed using the BDI. At subsequent visits (Visits 4, 6, and 8) change from baseline will be assessed using the TDI. General health status will be evaluated using the subject-completed EQ-5D questionnaire at Visits 2, 4, 6, and 8. Disease specific health status will be evaluated using the subject-completed St. George's Respiratory Questionnaire (SGRQ) at Visits 2, 4, 6, and 8, and the subject-completed COPD Assessment Test (CAT) at Visits 2, 6, and 8. The occurrence of adverse events will be evaluated throughout the study beginning at Visit 2. SAEs will be collected over the same time period as for AEs. However, any SAEs assessed as related to study participation (e.g., study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication, will be recorded from the time a subject consents to participate in the study up to and including any follow up contact. Additional safety assessments of vital signs (blood pressure and pulse rate), 12-lead ECGs and standard clinical laboratory tests (hematology and chemistry) will be obtained at selected clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* outpatient
* signed and dated written informed consent
* 40 years of age or older
* male and female subjects
* COPD diagnosis
* at least 10 pack-year smoking history
* post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and post-albuterol/salbutamol FEV1 of less than or equal to 70% predicted normal values
* score of greater than or equal to 2 on the Modified Medical Resarch Council Dyspnea Scale (mMRC)

Exclusion Criteria:

* women who are pregnant or lactating or are planning on becoming pregnant during the study
* current diagnosis of asthma
* other respiratory disorders other than COPD
* other diseases/abnormalities that are uncontrolled including cancer not in remission for at least 5 years
* chest x-ray or CT scan with clinically significant abnormalities not believed to be due to COPD
* hypersensitivity to anticholinergics, beta-agonists, lactose/milk protein or magnesium stearate or medical conditions associated with inhaled anticholinergics
* hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1
* lung volume reduction surgery within 12 months prior to Visit 1
* abnormal and clinically significant ECG at Visit 1
* significantly abnormal finding from laboratory tests at Visit 1
* unable to withhold albuterol/salbutamol at least 4 hours prior to spirometry at each visit
* use of depot corticosteroids within 12 weeks of Visit 1
* use of oral or parenteral corticosteroids, antibiotics for lower respiratory tract infection, or cytochrome P450 3A4 inhibitors, within 6 weeks of Visit 1
* use of long-acting beta-agonist (LABA)/inhaled corticosteroid (ICS) product if LABA/ICS therapy is discontinued withing 30 days of Visit 1
* use of ICS at a dose of >1000mcg/day of fluticasone propionate or equivalent within 30 days of Visit 1
* initiation or discontinuation of ICS within 30 days of Visit 1
* use of tiotropium or roflumilast within 14 days of Visit 1
* use of theophyllines, oral leukotriene inhibitors, long-acting oral beta-agonists, or inhaled long-acting beta-agonists within 48 hours of Visit 1
* short-acting oral beta-agonists within 12 hours of Visit 1
* use of LABA/ICS combination products only if discontinuing LABA therapy and switching to ICS monotherapy within 48 hours of Visit 1 for the LABA component
* use of sodium cromoglycate or nedocromil sodium within 24 hours of Visit 1
* use of inhaled short-acting beta-agonists, inhaled short-acting anticholinergics, or inhaled short-acting anticholinergic/short-acting beta-agonist combination products within 4 hours of Visit 1
* use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer)
* long-term oxygen therapy prescribed for >12 hours per day
* regular use of nebulized short-acting bronchodilators
* participation in acute phase of pulmonary rehabilitation program
* known or suspected history of alcohol or drug abse within 2 years prior to Visit 1
* anyone affiliated with the investigator site (e.g., investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member)
* previous exposure to GSK573719, GSK573719/GW642444 combination, GW642444 (vilanterol), or fluticasone furoate/GW642444 combination

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2011-03-01; Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (87):
- United States (19):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Phoenixville, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
- France (4):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Saint-Pierre
- Germany (12):
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (10):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Pietra Ligure (SV), Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Pisa, Tuscany
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Peru (8):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Jesus Maria, Lima region
  - GSK Investigational Site, San Borja, Lima region
  - GSK Investigational Site, San Isidro, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Santiago de Surco, Lima region
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Poland (7):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gidle
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubliniec
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Włocławek
  - GSK Investigational Site, Zabrze
- Romania (4):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (10):
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- Ukraine (9):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Maleki-Yazdi MR, Singh D, Anzueto A, Tombs L, Fahy WA, Naya I. Assessing Short-term Deterioration in Maintenance-naive Patients with COPD Receiving Umeclidinium/Vilanterol and Tiotropium: A Pooled Analysis of Three Randomized Trials. Adv Ther. 2017 Jan;33(12):2188-2199. doi: 10.1007/s12325-016-0430-6. Epub 2016 Oct 28. PMID 27796912
- [Derived] Decramer M, Anzueto A, Kerwin E, Kaelin T, Richard N, Crater G, Tabberer M, Harris S, Church A. Efficacy and safety of umeclidinium plus vilanterol versus tiotropium, vilanterol, or umeclidinium monotherapies over 24 weeks in patients with chronic obstructive pulmonary disease: results from two multicentre, blinded, randomised controlled trials. Lancet Respir Med. 2014 Jun;2(6):472-86. doi: 10.1016/S2213-2600(14)70065-7. Epub 2014 May 14. PMID 24835833
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113360 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening (Visit 1) completed a 7- to10-day run-in period and were then randomized to a 24-week treatment period. A total of 1141 par. were screened; 846 par. were randomized (3 par. were randomized [2 in error] and received no study drug) and 843 par. received at least one dose of study drug.
Groups:
- VI 25 µg: Participants received vilanterol (VI) 25 micrograms (µg) once daily (QD) via a dry powder inhaler (DPI). All participants also received placebo QD via a HandiHaler.
- UMEC/VI 62.5/25 µg: Participants received umeclidinium bromide (UMEC)/VI 62.5/25 µg QD via a DPI. All participants also received placebo QD via a HandiHaler.
- UMEC/VI 125/25 µg: Participants received UMEC/VI 125/25 µg QD via a DPI. All participants also received placebo QD via a HandiHaler.
- TIO 18 µg: Participants received tiotropium (TIO) 18 µg QD via a HandiHaler. All participants also received placebo QD via a DPI.
Period: Overall Study
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | TIO 18 µg
Started | 209 | 212 | 214 | 208
Completed | 165 | 181 | 173 | 177
Not Completed | 44 | 31 | 41 | 31
Not completed — Adverse Event | 10 | 10 | 15 | 9
Not completed — Lack of Efficacy | 17 | 9 | 5 | 7
Not completed — Protocol Violation | 7 | 1 | 4 | 0
Not completed — Protocol-defined Stopping Criteria | 2 | 3 | 10 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 7 | 8 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Tiotropium 18 µg: Participants received tiotropium (TIO) 18 µg QD via a HandiHaler. All participants also received placebo QD via a DPI.
- Total: Total of all reporting groups
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | Tiotropium 18 µg | Total
Number analyzed (Participants) | 209 | 212 | 214 | 208 | 843
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (9.10) | 63.0 (8.67) | 62.9 (8.87) | 62.6 (9.39) | 62.9 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 63 | 68 | 261
  Male | 143 | 148 | 151 | 140 | 582
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 3 | 7 | 9 | 6 | 25
  American Indian or Alaska Native | 19 | 16 | 21 | 20 | 76
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 0 | 1
  Asian - Japanese Heritage | 0 | 3 | 0 | 2 | 5
  White - White/Caucasian/European Heritage | 184 | 182 | 180 | 177 | 723
  Mixed Race | 3 | 4 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) on Day 169 (Week 24)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84, 112, 168, and 169. Baseline is defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after the previous morning's dosing (ie., trough FEV1 on Day 169 is the mean of the FEV1 values obtained 23 and 24 hours after the morning dosing on Day 168). Change from Baseline at a particular visit was calculated as the trough FEV1 at that visit minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline , smoking status, center group, day, and day by Baseline and day by treatment interactions. ITT=Intent-to-Treat; par.=participants. .
Time Frame: Baseline and Day 169
Population: ITT Population excluding par. from Investigator 040688: all randomized par. who received >=1 dose of study drug, except for those from Investigator 040688. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | TIO 18 µg
Number analyzed (Participants) | 162 | 177 | 167 | 173
Liters | 0.121 (0.0189) | 0.211 (0.0183) | 0.209 (0.0187) | 0.121 (0.0186)
Statistical Analysis 1: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.090, 95% CI 2-sided [0.039 to 0.142] — Least squares mean difference=UMEC/VI 62.5/25 µg minus VI 25 µg
Statistical Analysis 2: Comparison: UMEC/VI 62.5/25 µg vs TIO 18 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — nominal p-value; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.090, 95% CI 2-sided [0.039 to 0.141] — Least squares mean difference=UMEC/VI 62.5/25 µg minus Tio 18 µg
Statistical Analysis 3: Comparison: VI 25 µg vs UMEC/VI 125/25 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.088, 95% CI 2-sided [0.036 to 0.140] — Least squares mean difference=UMEC/VI 125/25 µg minus VI 25 µg
Statistical Analysis 4: Comparison: UMEC/VI 125/25 µg vs TIO 18 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.088, 95% CI 2-sided [0.036 to 0.140] — Least squares mean difference=UMEC/VI 125/25 µg minus TIO 18 µg

2. Secondary Outcome: Change From Baseline (BL) in Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Day 168
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1, 84, and Day 168 using the 0-6-hour post-dose FEV1 measurements collected on that day, which included pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits: 23 and 24 hours after the previous morning dose) and post-dose at 15 minutes, 30 minutes, 1 hour, 3 hours, and 6 hours. Change from BL at a particular visit was calculated as WM at that visit minus BL. Analysis was performed using a repeated measures model with covariates of treatment, BL (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), smoking status, center group, day, and day by BL and day by treatment interactions.
Time Frame: Baseline and Day 168
Population: ITT Population excluding participants from Investigator 040688. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | TIO 18 µg
Number analyzed (Participants) | 161 | 173 | 166 | 168
Liters | 0.178 (0.0189) | 0.254 (0.0183) | 0.263 (0.0187) | 0.181 (0.0187)

3. Other Pre Specified Outcome: Change From Baseline (BL) in the Mean Shortness of Breath With Daily Activities (SOBDA) Score for Week 24
Description: The newly developed SOBDA questionnaire assesses dyspnea or shortness of breath (SOB) with daily activities. The SOBDA questionnaire is made up of 13 items completed by the participant (par.) each evening prior to bedtime, when the par. is instructed to reflect on the current day's activities. The daily score is computed as the mean of the scores on the 13 items (>=7 items must have non-missing responses for this to be calculated). The par. is assigned a weekly mean SOBDA score ranging from 1 to 4 (greater scores indicate more severe breathlessness with daily activities) based on the mean of 7 days of data (>=4 of 7 days must be completed for a weekly mean to be calculated). Change from BL is the mean weekly SOBDA score minus BL. Analysis was performed using MMRM with covariates of treatment, BL (mean score in the week prior to treatment), smoking status, center group, week, week by BL and week by treatment interactions. This MMRM analysis only included Weeks 4, 8, 12, and 24.
Time Frame: Baseline and Week 24
Population: ITT Population excluding participants from Investigator 040688. Participants analyzed are those with data available at the presented time point; but, all participants without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | TIO 18 µg
Number analyzed (Participants) | 110 | 118 | 107 | 105
Scores on a scale | -0.16 (0.043) | -0.18 (0.042) | -0.18 (0.044) | -0.18 (0.044)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to 24 weeks).
Description: On-treatment SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | VI 25 µg | UMEC/VI 62.5/25 µg | UMEC/VI 125/25 µg | TIO 18 µg
Serious Adverse Events (participants affected / at risk) | 15/209 | 7/212 | 5/214 | 13/208
Other Adverse Events (participants affected / at risk) | 44/209 | 54/212 | 40/214 | 37/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VI 25 µg (N=209) | UMEC/VI 62.5/25 µg (N=212) | UMEC/VI 125/25 µg (N=214) | TIO 18 µg (N=208)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VI 25 µg (N=209) | UMEC/VI 62.5/25 µg (N=212) | UMEC/VI 125/25 µg (N=214) | TIO 18 µg (N=208)
Nasopharyngitis (Infections and infestations) | 17 | 21 | 14 | 16
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 7 | 8
Headache (Nervous system disorders) | 21 | 20 | 14 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 10 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.